CLINICAL TRIAL: NCT06678698
Title: Acute Effect of Photobiomodulation on Blood Pressure, Endothelial Function and Arterial Stiffness in Individuals with Hypertension: a Randomized Controlled Trial
Brief Title: Acute Effect of Photobiomodulation in Individuals with Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Lara Maria Bataglia Espósito, Physical Therapist, Master's student, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: UFSaoCarlosPBM
Record Dates: First submitted 2024-10-13; First posted 2024-11-07 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Hypertension
Keywords: hypertension; photobiomodulation; low-level light therapy
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Panel Group (Experimental): Participants who will receive full-body photobiomodulation irradiation, from a panel of LEDs
  Interventions: Device: Panel Effective Photobiomodulation Therapy
- Panel Sham Group (Sham Comparator): Participants who will receive full-body photobiomodulation irradiation, with the device turned-off
  Interventions: Device: Sham Panel Photobiomodulation Therapy
- Modified ILIB Group (Experimental): Participants who will receive photobiomodulation irradiation with the transcutaneous ILIB method
  Interventions: Device: Modified ILIB Photobiomodulation Therapy
- Modified ILIB Sham Group (Sham Comparator): Participants who will received photobiomodulation irradiation with the transcutaneous ILIB method, with the device turned-off
  Interventions: Device: Modified ILIB Sham Photobiomodulation Therapy

INTERVENTIONS:
Device: Panel Effective Photobiomodulation Therapy — Photobiomodulation therapy is the use of low-power light in biological tissues through a non-ionizing source of light (600 to 1.100 nm), with variable power between 1 and 500 mW and therapeutic goals.
  This group will receive photobiomodulation from a whole-body panel of low intensity LEDs
  Arms: Panel Group
Device: Sham Panel Photobiomodulation Therapy — Use of common red lamp to perform the sham photobiomodulation for the panel group
  Arms: Panel Sham Group
Device: Modified ILIB Sham Photobiomodulation Therapy — ILIB Therapy device turned off for the sham ILIB therapy
  Arms: Modified ILIB Sham Group
Device: Modified ILIB Photobiomodulation Therapy — Common laser used in ILIB mode for modified ILIB therapy
  Arms: Modified ILIB Group

SUMMARY:
This is a randomized, double-blind and sham-controlled clinical trial that aims to evaluate and compare the acute effect of full-body photobiomodulation (PBM) and modified ILIB (Intravascular laser irradiation of blood) on blood pressure, endothelial function and arterial stiffness in individuals with hypertension. Participants (n=48) will be equally, randomly and secretly allocated into one of 4 groups: Panel Group; Panel Sham Group; Modified ILIB group; and Modified ILIB Sham Group. Participants aged 40 to 60 years old, diagnosed with hypertension and using control drugs for at least 3 months will be included. Participants will be assessed at pre- and post-intervention for: BP; endothelial function; arterial stiffness; blood nitrite; and thermography. In the post-intervention period, the ambulatory blood pressure monitoring will also be carried out. Participants will receive a single application of PBM, which, depending on the group, may be full-body irradiation from an LED panel (660 nm; 25.34 J/cm²; 42.24 mW/cm²), modified ILIB (660 nm; 42,462 J/cm²; 35.385 W/cm²), or the respective sham therapies. Data homogeneity and normality will be verified by the Levene and Shapiro-Wilk tests, which will determine the choice of subsequent tests. A statistical significance of 5% will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary or irregularly inactive individuals (IPAQ)
* Both sexes
* Age between 40 to 60 years old
* Clinical diagnosis of hypertension for at least 3 months with difficulty in blood pressure control
* Hypertension classification up to stage 2
* Individuals who have a prescription for hypertension control drugs and have been using these drugs for at least 3 months

Exclusion Criteria:

* Diabetes diagnosis
* Smokers
* BMI > 30 kg/m²
* Cardiac pacemaker use
* Presence of arrhythmias or other decompensated cardiovascular diseases
* Musculoskeletal, orthopedic or neurological conditions that make it unable to participate in the procedures
* Presence of cognitive deficits that make it difficult to understand the assessments
* Presence of active neoplasia, under suspicion or after 5 years in remission period
* Presence of tattoos (covering a large body area, or the anterior wrist region)
* Photosensitive drugs use
* Pregnant women or under suspicion
* Presence of epilepsy or seizures
* Participants who present a systolic blood pressure ≥ 180 mmHg and/or diastolic blood pressure ≥ 110 mmHg on the day of the intervention

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Diastolic Blood Pressure | Acute effect (immediately post-intervention until 24 hours after)
  Diastolic blood pressure measured in millimeters of mercury (mmHg)

SECONDARY OUTCOMES:
Systolic Blood Pressure | Acute effect (immediately post-intervention until 24 hours after)
  systolic blood pressure measured in millimeters of mercury (mmHg)
Mean Arterial Pressure | Acute effect (immediately post-intervention until 24 hours after)
  mean arterial pressure measured in millimeters of mercury (mmHg)
Endothelial Function | Acute effect (About 25 minutes post-intervention)
  Endothelial function measured by flow-mediated dilation, with a brachial artery ultrasound
Arterial Stiffness | Acute effect (About 15 minutes post-intervention)
  Arterial stiffness measured by pulse wave velocity
Blood Nitrite | Acute effect (1 hour post-intervention)
  Blood nitrite levels

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of São Carlos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No